CLINICAL TRIAL: NCT03406923
Title: Self-efficacy, Beliefs and Adherence- Pilot and Feasibility Trial of a Pharmacist-led Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); William S. Middleton Memorial Veterans Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017-0951; Protocol Version 3/27/2020 (Other: UW Madison); A561000 (Other: UW Madison); PHARM/PHARMACY (Other: UW Madison)
Record Dates: First submitted 2017-12-28; First posted 2018-01-23 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus
Keywords: Health literacy; Self-efficacy; Beliefs about diabetes; Beliefs in medicines
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Receive usual care only.
- Health literacy-psychosocial support (Experimental): Receive 6-week sessions of individual health literacy-psychosocial support in addition to usual care. The health literacy-psychosocial support intervention includes 45-minute face-to-face counseling at week 1 and week 6 as well as weekly phone calls (week 2 to week 5.)
  Interventions: Other: Health literacy-psychosocial support

INTERVENTIONS:
Other: Health literacy-psychosocial support — The intervention is based upon enhancing patient health literacy-related attributes by (1) addressing the barriers to patients' self-efficacy by working with the patient to minimize the barriers (2) clarifying the patient beliefs about diabetes and diabetes medications, and (3) developing personalized action plans. We will tailor the intervention to each patient, so, the details of the content of each session will depend on the individual's self-efficacy, beliefs in illness and medicines, and health literacy level obtained at baseline. In addition to the 45-minute scheduled sessions, patients will be able to call the clinical pharmacist on the phone during the 6-week session at their discretion, for patient-driven support for self-management of goals and skills.
  Arms: Health literacy-psychosocial support

SUMMARY:
This study uses an intervention mixed methods design. The overall purpose is to improve medication adherence and assess the clinical impact on diabetes outcomes among patients with uncontrolled diabetes. We will examine if usual care combined with a clinic-based health literacy/psychosocial support intervention improves medication adherence compared to usual care alone. A randomized controlled trial will be conducted at William S. Middleton Memorial Veterans Hospital in Madison, targeting individuals with uncontrolled diabetes. The patient-centered health literacy intervention will focus on enhancing patients' self-efficacy and addressing patients' negative beliefs in medicine and illness.

DETAILED DESCRIPTION:
The study will improve medication adherence for patients with diabetes using two strategies: 1) addressing health literacy by reducing the complexity of diabetes content disseminated to patients during medication counseling and 2) addressing health literacy by enhancing patient-pharmacist communication. The second strategy aims to improve the psychosocial support offered to patients by building self-efficacy and addressing negative beliefs about medicines and diabetes. Together, the patient and the pharmacist can work together towards goal setting, problem solving, and negotiation of competing priorities.

Currently, with usual care, the pharmacist confirms if patients understand how to take medications correctly, adjusts diabetes medications, and monitor patients' hemoglobin A1C levels periodically to make sure that patients are capable of managing their diabetes appropriately. With the proposed intervention, the pharmacist will identify patients' concerns and barriers to medication taking and self-care with diabetes with an emphasis on self-efficacy, negative beliefs in medicine and illness. Then the pharmacist will provide individualized plans and set specific goals with each patient by strengthening their confidence in medication use and health literacy skills in navigating health information for diabetes self-care. The methods described for the intervention are in line with the current clinic workflow and will not require a substantial change to the current system for counseling diabetes patients. Knowledge change often does not lead to behavior change. Hence, the intervention will innovatively focus on moving knowledge towards action as the clinical pharmacist works with patients in assessing health literacy, identifying their barriers to medication use, including lack of self-efficacy, addressing negative beliefs about diabetes and diabetes medications; towards problem solving, and developing goals and action plans that will improve medication adherence and glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking men and women 18-80 years old with diabetes
* Taking oral diabetes medications and/or insulin
* One hemoglobin A1C measure of 8% or greater in the last 18 months
* A score less than 25 on the Medication Adherence Rating Scale (MARS-5)

Exclusion Criteria:

* Unable to provide informed consent
* Younger than 18 years old or older than 80 years old
* Unable to understand English
* Do not take oral diabetes medications and/or insulin
* A score equal to 25 on the Medication Adherence Rating Scale (MARS-5)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in diabetes medication adherence | Baseline, 3 months, and 6 months after the intervention
  Proportion of days covered and the 5-item Medication Adherence Rating Scale (MARS-5) will be used to measure diabetes medication adherence. The minimum score for the MAR scale is 5 and the maximum score is 25. Total score ranges from 5-25; Higher scores represent higher self-reported adherence.
Change in diabetes control | Baseline and 6 months after the intervention
  Hemoglobin A1c will be abstracted from electronic medical records using the most recent value for each participant within the prior six months.

SECONDARY OUTCOMES:
Self-efficacy for medication use | Baseline, 6 weeks, and 3 months after the intervention
  Self-efficacy for medication use will be measured using the 13-item Self-efficacy for Appropriate Medication Use Scale. The minimum score is 13 and the maximum score is 39. Higher scores represent higher confidence in adhering to medication use.
Illness beliefs | Baseline, 6 weeks, and 3 months after the intervention
  Illness beliefs will be measured using the 9-item the Brief Illness Perception Questionnaire. A higher score indicates a more threatening view of the illness. Total score ranges from 0-80.
Beliefs in medicines | Baseline, 6 weeks, and 3 months after the intervention
  Beliefs in medicines will be measured using the 10-item Belief about Medicines Questionnaire. The 10-item Belief about Medicines Questionnaire (BMQ) has the necessity beliefs and concern beliefs sub-scale (five items each). The scale has five-point Likert-type responses ranging from strongly disagree to strongly agree. Each sub-scale has scores ranging from 5-25, with a higher score meaning stronger concern or necessity beliefs about the medicine.
Health literacy | Baseline and 6 months after the intervention
  Health literacy will be measured using the 6-item Newest Vital Sign. Each question will be scored "0" for incorrect and "1" for correct yielding a total score ranging from 0 to 6, with higher scores indicating better health literacy. Scores less than 2 represented a high likelihood (50% or more) of limited (inadequate) health literacy, 2 to 3 indicated the possibility of limited (marginal) health literacy, and more than 3 suggested adequate health literacy.
Experiences and perceptions of the intervention processes and outcomes | 6 months after the intervention
  A phenomenological qualitative approach using semi-structured 60-minute in-depth interviews will be conducted with 15 intervention participants.

CONTACTS AND LOCATIONS:
Overall Officials: Olayinka Shiyanbola, PhD, BPharm, Principal Investigator — School of Pharmacy, University of Wisconsin, Madison
Locations (1):
- William S. Middleton Memorial Veterans Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farmer KC. Methods for measuring and monitoring medication regimen adherence in clinical trials and clinical practice. Clin Ther. 1999 Jun;21(6):1074-90; discussion 1073. doi: 10.1016/S0149-2918(99)80026-5. PMID 10440628
- [Background] Keogh KM, Smith SM, White P, McGilloway S, Kelly A, Gibney J, O'Dowd T. Psychological family intervention for poorly controlled type 2 diabetes. Am J Manag Care. 2011 Feb;17(2):105-13. PMID 21473660
- [Background] Lee YJ, Shin SJ, Wang RH, Lin KD, Lee YL, Wang YH. Pathways of empowerment perceptions, health literacy, self-efficacy, and self-care behaviors to glycemic control in patients with type 2 diabetes mellitus. Patient Educ Couns. 2016 Feb;99(2):287-94. doi: 10.1016/j.pec.2015.08.021. Epub 2015 Sep 2. PMID 26341940
- [Background] Unni E, Shiyanbola OO, Farris KB. Change in Medication Adherence and Beliefs in Medicines Over Time in Older Adults. Glob J Health Sci. 2015 Sep 1;8(5):39-47. doi: 10.5539/gjhs.v8n5p39. PMID 26652095
- [Background] Shiyanbola OO, Farris KB, Chrischilles E. Concern beliefs in medications: changes over time and medication use factors related to a change in beliefs. Res Social Adm Pharm. 2013 Jul-Aug;9(4):446-57. doi: 10.1016/j.sapharm.2012.07.003. Epub 2012 Sep 19. PMID 22999805